CLINICAL TRIAL: NCT03387475
Title: Phase II Trial Evaluating Low-dose Deferasirox (DFX) in Patients With Low-risk (MDS) Myelodysplastic Syndrome Resistant or Relapsing After ESA Agents (LODEFI)
Brief Title: Evaluating Low-dose Deferasirox (DFX) in Patients With Low-risk MDS Resistant or Relapsing After ESA Agents
Acronym: LODEFI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.064
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Myelodysplasia
Keywords: efficacy; safety
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox (Experimental): efficacy of 3.5mg/kg/day
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — iron chelation
  Other Names: exjade

SUMMARY:
Patients with low-risk MDS verifying the eligibility criteria may be included in the study.

DETAILED DESCRIPTION:
Patients will receive the number of DFX tablets (Exjade, cp film-coated, 90mg or 360mg), in relation to their body weight to be closer to 3.5mg / kg / d for 12 months.

At one month and six months of treatment, the residual plasma levels of DFX will be measured in patients (sent to the Bordeaux laboratory of Biochemistry, Pr Molimard) to allow the dosage to be adjusted (plasma objective of 3 μM).

At inclusion (J1) and at 6 months of treatment, a dosage of NTBI and hepcidine will be performed.

If patients become transfusion-dependent (≥) 2 packed red cells (RBP) per 2-month period evaluated over 6 months, they will stop low-dose DFX and go out of protocol to receive DFX at 20mg / kg (according to EMEA authorization) for iron chelation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS according to WHO 2008 criteria (refractory anemia with multilineage dysplasia, RA (refractory anemia), refractory anemia with ringed sideroblasts (RARS) including CMML-1 (chronic myelomonocytic leukemia) type 1 with <10% blasts)
2. low risk (IPSS-R very low, low and intermediate)
3. in primary or secondary failure after erythropoiesis stimulating agents (ESAs), (either epoetins (≥60,000 units / week), or darbepoetin (≥250 μg / week), administered for at least 12 weeks, as defined by the IWG criteria 2006 (no erythroid response at 12 weeks, or more than 15g / l decrease in Hb after response to ESAs) PS: Patients with low transfusion of less than (<) 4RBP assessed over 4 months (RBP administered for patients with Hb ≤ 9g / dl) will be accepted)
4. age ≥ 18 years
5. ECOG ≤2
6. informed consent dated and signed
7. affiliated to a social security scheme
8. Women and men of childbearing potential must have effective contraception throughout the duration of the study and up to 4 days after the last administration of deferasirox

Exclusion Criteria:

1. Transfusion dependent patient (≥) 2 red blood cells (RBP) per 2-month period evaluated over 4 months between M-4 and M0
2. Patients with high-risk MDS (based on IPSS-R) and patients with other hematologic and non-haematological malignancies who should not benefit from chelation therapy due to rapid progression of their disease
3. Ferritin <200 ng / ml
4. Iron overload: ferritin> 1000 ng / ml
5. Creatinine clearance according to MDRD ≤60 ml / min
6. 5q- deletion to karyotype
7. Patient eligible for allograft
8. Patient participating in another interventional clinical study or exclusion period from another study
9. History of cancer treated or untreated for less than 5 years, whether or not there are signs of relapse or metastases, with the exception of basocellular cancers.
10. Persons referred to in Articles L1121-5 to L1121-8 of the CSP: pregnant woman, parturient, mother who is breastfeeding, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure, can not not be included in clinical trials.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients without transfusion-dependence at 12 months. | 12 months
  Percentage of patients without transfusion-dependence at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Park, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de GRENOBLE ALPES, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
e crf